CLINICAL TRIAL: NCT07078630
Title: Co-supplementation of Ferrous Iron With Formulated Curcumin Reduces Hepcidin Response in Trained Individuals: a Cross-over, Double-blinded, Placebo-controlled Human Intervention Study
Brief Title: Modulation of hepcidIN With Co-supplementation of Iron and FORMulated Curcumin in Recreational Athletes
Acronym: IN-FORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: Pharmako Biotechnologies Pty Ltd (Unknown)
Responsible Party: Principal Investigator, Mohammed Gulrez Zariwala, Professor of Translational Physiology, University of Westminster
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ETH2223-1363
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Iron Supplementation and Gastrointestinal Health; Iron Deficiency
Keywords: Iron; Ferrous sulphate; Curcumin; IFABP; Ferritin; Interleukin-6; Hepcidin; Iron deficiency; Anaemia; Inflammation; Oxidative stress; Supplement; Gastrointestinal symptoms; Nutraceutical
MeSH Terms: conditions — Iron Deficiencies; Anemia; Inflammation | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomised, placebo-controlled, crossover.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous iron + placebo (Placebo Comparator): * Dried ferrous sulphate tablet, 200mg providing 65 mg of elemental iron (Remedy Healthcare, UK).
  * Placebo capsule containing maltodextrin and a food grade dye (yellow 5 or E102) (Fast Colours LLP, Huddersfield, UK)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Ferrous sulphate 200mg oral tablet providing 65 mg of elemental iron
- Ferrous iron + HydroCurc (Active Comparator): * Dried ferrous sulphate, 200mg tablet providing 65 mg of elemental iron (Remedy Healthcare, UK).
  * HydroCurc (Gencor Pacific Limited, Lantau Island, Hong Kong), 500 mg capsule containing not less than 90% 115 curcuminoids (85% curcumin), formulated in 10% LipiSperse® (Pharmako Biotechnologies Pty Ltd, 116 Sydney, Australia), a delivery system comprising a proprietary mixture of surfactants, polar lipids 117 and solvents.
  Interventions: Dietary Supplement: HydroCurc®; Dietary Supplement: Ferrous sulphate 200mg oral tablet providing 65 mg of elemental iron

INTERVENTIONS:
Dietary Supplement: Placebo — Participants instructed to intake the placebo capsule along with the ferrous sulphate tablet, separated from food, tea or coffee, at the same time of the day.
  Arms: Ferrous iron + placebo
Dietary Supplement: HydroCurc® — Participants instructed to intake the HydroCurc® capsule along with the ferrous sulphate tablet, separated from food, tea or coffee, at the same time of the day.
  Arms: Ferrous iron + HydroCurc
Dietary Supplement: Ferrous sulphate 200mg oral tablet providing 65 mg of elemental iron — Participants instructed to intake the ferrous sulphate tablet along with the HydroCurc® or the placebo together, preferably and separated from food, tea or coffee, at the same time of the day.

SUMMARY:
Iron deficiency and iron deficiency anaemia are common among endurance athletes partly due to a repeated post-exercise elevation of hepcidin, a hormone limiting iron entry through the intestine. Oral iron supplementation also causes stimulation of hepcidin that adds on to the exercise-intrinsic stimulation of this hormone further reducing iron absorption. Both oral ferrous iron therapy and performance running are known to cause undesired gastrointestinal symptoms. Curcumin, a polyphenol from turmeric, has been previously shown to reduce hepcidin levels in resting individuals and to protect the gastrointestinal (GI) function but its effect on active individuals supplementing with iron remains unclarified.

The objective of this research study is to learn about the effects of a formulated curcumin (HydroCurc®) on intestinal health and regulation mechanisms of body iron levels in recreationally active athletes supplementing with iron.

The main questions to answer are:

Does HydroCurc® influence iron regulatory mechanisms in resting conditions? Does HydroCurc® influence iron regulatory mechanisms in post-exercise conditions? Does HydroCurc® alleviate iron supplementation- and exercise-related gastrointestinal adverse events

Researchers will compare HydroCurc® to a placebo (a look-alike substance that contains no drug) to see if there are any significant changes.

Participants will:

* Perform a fitness test
* Take iron and HydroCurc for seven days
* Complete questionnaires on their gastrointestinal health
* Complete anthropometric testing
* Undergo blood sampling

DETAILED DESCRIPTION:
Intervention study with two treatment groups in a randomised, double-blinded, placebo-controlled, crossover design.

Healthy recreationally active athletes will perform a VO2 max test to determine their aerobic capacity. A blood sample will be taken prior to the test as baseline measurement. Following treatment with iron plus either HydroCurc or a matched placebo for a week, participants will run on a treadmill for one hour at 70% of their maximal capacity. Blood samples will be collected before, immediately after, one hour post- and three hours post-exercise. Gastrointestinal symptoms will be assessed via validated questionnaires during the supplementation period and the experimental visits. All participants will observe a minimum of a two-week washout period. All participants will attend visits fasting for a minimum of four hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-40 years) endurance male & female runners.
* All participants will be accustomed to exercising at least 150 minutes per week, meeting the minimum NHS exercise recommendation.
* Participants will be fit enough to run for 60 minutes on a treadmill at 70% of their V̇O2max. To that end, participants will undergo a fitness test in the screening visit.

Exclusion Criteria:

* <18 years or >40 years
* Those with deficient/excess/abnormal iron levels according to UK guidelines &/or haemochromatosis
* Any allergies/health issues related to items being ingested.
* Any illnesses or those on medication
* Those on iron or curcumin supplements
* Any pregnant or lactating women
* Any women who are trying to conceive
* Any gastrointestinal disorders
* Any eating disorders
* Any abnormal blood pressure levels
* Consumption of >14 units of alcohol/week
* Devices such as pacemakers
* Smokers
* Renal disorders
* Dieters

These criteria will be self-reported.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Concentration of iron absorption regulatory hormone in athletes supplementing with ferrous iron in resting conditions | Hepcidin measured 1 day post supplementation
  Hepcidin, ng/mL
Exercise-associated hepcidin concentration in athletes supplementing with ferrous iron | Hepcidin measured 180 minutes post-exercise
  Hepcidin, ng/mL
Ferrous iron-associated iron status in athletes | Ferritin measured 1 day post supplementation
  Ferritin, ng/mL
Change of exercise-associated inflammation in ferrous iron supplemented athletes | Interleukin-6 measured 0- and 60-minutes post-exercise
  Interleukin-6, pg/mL

SECONDARY OUTCOMES:
Exercise-associated intestinal damage in ferrous iron supplemented athletes | IFABP measured 0- and 60-minutes post-exercise
  Intestinal Fatty Acid Binding Protein (IFABP), pg/mL
Incidence and frequency of ferrous iron associated-gastrointestinal symptoms | Gastrointestinal symptoms analysed daily throughout the supplementation period (seven continuous days)
  Subjective analysis via Oral Iron Supplement Questionnaire
Number of participants supplementing with ferrous iron and reporting exercise-associated gastrointestinal symptoms | Gastrointestinal symptoms measured 30 minutes after the commencement of the exercise, 0-, 60- and 180- minutes post-exercise.
  Subjective analysis via gastrointestinal symptom questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed G Zariwala, PhD, Principal Investigator — University of Westminster
Locations (1):
- University of Westminster London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Szymanski MC, Gillum TL, Gould LM, Morin DS, Kuennen MR. Short-term dietary curcumin supplementation reduces gastrointestinal barrier damage and physiological strain responses during exertional heat stress. J Appl Physiol (1985). 2018 Feb 1;124(2):330-340. doi: 10.1152/japplphysiol.00515.2017. Epub 2017 Sep 21. PMID 28935827
- [Background] Peters HP, Bos M, Seebregts L, Akkermans LM, van Berge Henegouwen GP, Bol E, Mosterd WL, de Vries WR. Gastrointestinal symptoms in long-distance runners, cyclists, and triathletes: prevalence, medication, and etiology. Am J Gastroenterol. 1999 Jun;94(6):1570-81. doi: 10.1111/j.1572-0241.1999.01147.x. PMID 10364027
- [Background] Ishibashi A, Maeda N, Kamei A, Goto K. Iron Supplementation during Three Consecutive Days of Endurance Training Augmented Hepcidin Levels. Nutrients. 2017 Jul 30;9(8):820. doi: 10.3390/nu9080820. PMID 28758951
- [Background] Laine F, Laviolle B, Bardou-Jacquet E, Fatih N, Jezequel C, Collet N, Ropert M, Morcet J, Hamon C, Reymann JM, Loreal O. Curcuma decreases serum hepcidin levels in healthy volunteers: a placebo-controlled, randomized, double-blind, cross-over study. Fundam Clin Pharmacol. 2017 Oct;31(5):567-573. doi: 10.1111/fcp.12288. Epub 2017 May 7. PMID 28370178
- [Background] Larsuphrom P, Latunde-Dada GO. Association of Serum Hepcidin Levels with Aerobic and Resistance Exercise: A Systematic Review. Nutrients. 2021 Jan 27;13(2):393. doi: 10.3390/nu13020393. PMID 33513924
- [Background] Keller K, Friedrich O, Treiber J, Quermann A, Friedmann-Bette B. Iron deficiency in athletes: Prevalence and impact on VO2 peak. Nutrition. 2024 Oct;126:112516. doi: 10.1016/j.nut.2024.112516. Epub 2024 Jun 10. PMID 39002373